CLINICAL TRIAL: NCT04690803
Title: The Effect of Cooling on Sclerotherapy Efficacy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Goldman, Butterwick, Fitzpatrick and Groff (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: ScleroTT2019-01
Record Dates: First submitted 2020-12-28; First posted 2020-12-31 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Leg Veins

STUDY DESIGN:
Intervention Model Description: sclerotherapy with forced-air cooling during treatment.
Who Masked: Investigator
Masking Description: evaluator-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- treatment with forced-air cooling (Active Comparator): comparing treatment with and without forced-air cooling in a comparative lower extremity model
  Interventions: Drug: air cooling
- treatment without forced-air cooling (No Intervention): comparing treatment without forced-air cooling in a comparative lower extremity model

INTERVENTIONS:
Drug: air cooling — intervention is adding air-cooling to treatment
  Arms: treatment with forced-air cooling

SUMMARY:
The primary objective of this study is to evaluate the efficacy of sclerotherapy with forced-air cooling during treatment.

DETAILED DESCRIPTION:
Study Objective: The primary objective of this study is to evaluate the efficacy of sclerotherapy with forced-air cooling during treatment.

Study Design: This will be an investigator-initiated, evaluator-blinded, randomized-controlled, prospective, single-center clinical trial.

Study Population: 20 evaluable subjects with bilateral lower extremity reticular and telangiectatic veins, who meet all study inclusion/exclusion criteria will be considered for entry into the study.

ELIGIBILITY:
Inclusion Criteria:

* The subject is a male or female of skin type I to IV between 25 and 75 years of age.
* The subject has mild venous disease (CEAP Class C1) (CLINICAL SEVERITY ETIOLOGY OR CAUSE ANATOMY AND PATHOPHYSIOLOGY)
* Reticular veins and telangiectasias on symmetrical bilateral lower extremities.
* The subject is willing to follow study instructions and complete all required visits, as well as has agreed to and signed the written informed consent form.
* The subject is healthy as judged by medical history and investigator's assessment of current health.
* The subject is not suffering from any skin condition (infection, dermatosis, etc.) that in the opinion of the investigator may place them at risk.
* Females of childbearing potential must use one of the following types of birth control for the duration of the study. These include: Oral contraceptives, contraceptive patches/rings/implants, Implanon®, Depo-Provera®, double-barrier methods (e.g. condoms with spermicide), abstinence, or partner vasectomy, with a documented second acceptable method of birth control should they become sexually active. All birth control measures must be in consistent use for at least 30 days prior to the start of study.

Exclusion Criteria:

* A subject requires greater than 10 mL total of glycerin, including a maximum of 6 mL of polidocanol for foam sclerotherapy, for either lower extremity during a single leg treatment.
* Asymmetric amount, distribution, and/or severity of reticular veins and/or telangiectasias between lower extremities
* The subject has a CEAP Class of C2 or greater, as evidenced by clinically apparent varicosities, venous stasis, stasis dermatitis, lipodermatosclerosis, and/or venous ulceration (or history of lower leg ulcerations).
* The subject has history of or current great saphenous vein (GSV), saphenofemoral junction (SFJ), or saphenopopliteal junction (SPJ) incompetency based on prior Doppler and/or duplex evaluation or has physical exam findings suspicious for it.
* The subject has a history of deep vein thrombosis, thrombophlebitis, thromboembolic disease, and/or underlying hypercoagulable medical condition (e.g. hemophilia, Factor V deficiency).
* The subject has a history of uncontrolled or severe asthma, or asthma requiring hospitalization or intubation.
* The subject has a history of allergic reactions to sclerosing agent.
* The subject has a history of allergic reaction or sensitivity to lidocaine or epinephrine.
* Any of the following medications, procedures or treatments to the purposed treatment area/s

  1. Within 6 months prior to screening visit (i.) The subject has undergone sclerotherapy
  2. Within 3 months prior to screening visit (I.) NO OTHER COSMETIC OR SURGICAL TREATMENTS TO THE PURPOSED TREATMENT AREA/S
* The subject is non-ambulatory or poorly ambulatory.
* The subject has a history of neurological conditions.
* The subject is pregnant, lactating, or in child bearing age (and sexually active) and not using an approved contraceptive measure.
* The subject is taking disulfiram, tamoxifen, or oral hormone therapy (not including hormonal birth control).
* The subject has a history of noncompliance with clinical protocols.
* The subject has participated in any other clinical trial that involves an investigational medication or device within the last 30 days.
* Planning to have any treatments or procedures to bilateral lower extremities for the duration of the trial.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-01-06 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
to evaluate the effect of forced-air cooling on sclerotherapy | 1 year
  to evaluate the effect of forced-air cooling on sclerotherapy of lower extremity telangiectasias and reticular veins. This will be assessed by comparing treatment with and without forced-air cooling in a comparative lower extremity model.

SECONDARY OUTCOMES:
is to compare reticular vein and telangiectasia diameter measurements | 1 year
  to compare reticular vein and telangiectasia diameter measurements via a polarized LED wireless digital microscope before treatment and during cooling in the forced-air cooling group.

CONTACTS AND LOCATIONS:
Locations (1):
- West Dermatology Research Center/Cosmetic Laser Dermatology, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No